CLINICAL TRIAL: NCT01102959
Title: The Effectiveness of Photographic Educational Material on Carbohydrate Counting for Adolescents With Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sandra Josefina Ferraz Ellero Grisi, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1182/07
Record Dates: First submitted 2010-04-07; First posted 2010-04-13 (Estimated); Last update posted 2010-04-13 (Estimated); Status verified 2010-03

CONDITIONS: Diabetes Mellitus
Keywords: EDUCATION; DIABETES MELLITUS; ADOLESCENT; DIABETIC DIET
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Photographic Material (Experimental): Photographic Educational Material on Carbohydrate Counting
  Interventions: Device: Photographic Educational Material

INTERVENTIONS:
Device: Photographic Educational Material — Photographic Educational Material on Carbohydrate Counting
  Other Names: Photo; Education; Nutrition

SUMMARY:
The hypothesis of this study focuses on obtaining accurate information on the effectiveness of photographic educational material on orientation of carbohydrate counting for adolescents with diabetes.

DETAILED DESCRIPTION:
The adolescents with diabetes at the Pediatric Endocrinology and Diabetes outpatient clinic, will be randomly distributed between two groups: those who will receive orientation on carbohydrate counting through photographic educational material and those through a list of foods equivalent.

Research will follow 3 steps:

First, data will be collected on age, gender, BMI, HbA1C, schooling, type of educational material and parents grade level; answer sheets will be applied to evaluate previous knowledge on carbohydrate counting; orientation will be provided on counting with photo material or list.

Second, after a month of using the educational material, a quiz by phone will be conducted with the sole intent to reinforce orientation.

Third, two days later, adolescents will be directed to the experimental kitchen to see portions of real food and provide answers on amount or choice of carbohydrate.

Statistical tools will be applied to evaluate results.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents with diabetes aged 11 years to 19 years who count carbohydrates in their diet.
* Adolescents with more than 6 years of study .
* There is no restriction ethnic, social, gender, nutrition status, type of diabetes.

Exclusion Criteria:

* Adolescents with diabetes aged 11 years to 19 years who not count carbohydrate counting in your diet.
* Adolescents with less than 6 years of study.
* Adolescents who don't want to participated in this research.

Ages: 11 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Number the answers correct or incorrect on carbohydrate counting in portions of real food | 1 month
  One month after intervention the adolescents' ability in CH counting will be tested.
  In an experimental kitchen, the adolescents will look at portions of real food and will provide answer sheet on carbohydrate counting.
  The answer sheet have 11 questions based on the different food groups, each group will be represented by one type of food.
  We will compare of photographic education material and list of foods equivalent by analysis of the answering sheets.
  We will categorize the answers by correct or incorrect. The statistics analysis we will compare the average score of each group.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre A. Ferraro, Phd, Study Chair — University of São Paulo General Hospital
Locations (1):
- University of São Paulo General Hospital, São Paulo, São Paulo, Brazil